CLINICAL TRIAL: NCT02587091
Title: Effectiveness of Advertising Availability of Prenatal Ultrasound on Uptake of Antenatal Care in Rural Uganda: a Randomized Trial
Brief Title: Effectiveness of Advertising Availability of Prenatal Ultrasound on Uptake of Antenatal Care in Rural Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bridge to Health Medical and Dental (Other)
Collaborators: Kigezi Healthcare Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Antenatal Care; Maternal Health

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control Arm (No Intervention): In this arm communities were told by word of mouth advertisement that a comprehensive antenatal care clinic would be held. There was no advertisement of portable ultrasound.
- Intervention Arm (Experimental): In this arm communities were told by word of mouth advertisement that a comprehensive antenatal care clinic would be held. In addition, it was advertised that portable ultrasound would be provided free of charge in addition to standard comprehensive antenatal care.
  Interventions: Behavioral: Portable obstetric ultrasound

INTERVENTIONS:
Behavioral: Portable obstetric ultrasound — This intervention was advertised at the cluster level
  Arms: Intervention Arm

SUMMARY:
A cluster randomized trial was conducted across eight rural sub-counties in southwestern Uganda. This study was conducted to determine the impact of advertising free obstetric ultrasound on the attendance to antenatal care clinics.

DETAILED DESCRIPTION:
Study Design We conducted a non-blinded cluster-randomized controlled trial to evaluate the effectiveness of advertising prenatal portable obstetric ultrasound (pOBU) on uptake of antenatal care (ANC) services. This study design was selected to mitigate confounding variables and use the natural landscape of the region (described below), which is conveniently divided into geographically isolated but otherwise homogenous sub-counties, to our advantage.

The study was conducted in Kabale District, a rural highland located in southwestern Uganda. It is roughly 560 km from the capital city of Kampala and has a population of approximately 522,000. It is divided into three regions - north, central and south, and is further subdivided into 22 sub-counties, with 11 in the North, four centrally and seven in the South.

Ethics approval was obtained from Lakeridge Health Corporation in the city of Oshawa, Canada as well as Mbarara University of Science and Technology (MUST) in Mbarara, Uganda. The study protocol can be found at the following link:

http://bridgetohealth.ca/study-protocol/

Study Population All sub-counties of southern and northern regions of Kabale district were eligible for inclusion as a cluster in this study. This population predominantly engages in subsistence agriculture. There is very limited data describing the healthcare of this rural and isolated region, and it is believed that government statistics are often inaccurate. The Ugandan Ministry of Health, numerous non governmental organizations (NGOs) and other faith-based organizations provide for the regions' healthcare. Data suggests that uptake of any ANC services is close to 66%, with only one third of these women returning for a fourth visit or delivering in a healthcare facility (HCF).

All women who were currently aware of being pregnant and presented to ANC were eligible for inclusion into the study. No pregnant woman who presented to clinic was excluded from the study. All patients provided written informed consent on a form developed in collaboration with the MUST ethics board. Many patients were illiterate or unable to read the consent form as it was written in English. A bilingual Ugandan midwife, translated the consent form and verbally explained its contents for each patient as they were checked into the clinic. It was clearly stated that any patient who chose to not engage in the research study would still receive full ANC care.

Randomisation and Masking Twenty-two sub-counties were assessed for inclusion, of these 18 were randomised to the intervention (n=4) or control group (n=4). The four sub-counties in the central region were intentionally excluded from the study design because they are primarily composed of urban and sub-urban communities and effectively divide the northern and southern regions. Four control sites (sub-counties) were randomly selected from the southern wing and four intervention sites were randomly selected from the northern wing. Selection of northern versus southern counties for intervention or control groups, as well as selection of which subcounties within each region and in which order they would be visited was all selected at random. Random selection was conducted by the statisticians at MUST using a simple random number program in MS-Excel.

All eight sub-counties in the control and treatment arm received advertisement by word of mouth (WOM) regarding ANC. The control arm received no advertisement of pOBU. When consent was obtained in the control arm there was intentional masking of pOBU. Following completion of initial consent and an entrance survey all women were provided with a debriefing form explaining the presence of ultrasound, including communities where it had not been advertised, and again consent was obtained to participate in the research study. Any women who chose to not engage in the research study were provided with complete ANC services, including pOBU.

Communities were randomly selected as stated above to receive messaging of pOBU. However, the control communities were chosen to be visited en bloc in the first four days, as opposed to alternating control then intervention on each day. This was done specifically to avoid contamination with radio messaging of pOBU, which was felt to possibly cross geographic boundaries. Sunday was intentionally avoided as a study day as most patients in the population ascribe to the Catholic faith and would not attend any clinics if held on that particular day.

Intervention The intervention itself was advertising the availability of clinic and pOBU at the cluster level (sub-county). The initial study design had only two groups as described above in randomisation. However, the protocol was amended during the study due to interim analysis results demonstrating WOM advertising of pOBU was not successful in increasing uptake of ANC. It was hypothesized that the population was unable to spread this message as many did not know what pOBU was, and therefore could not relay the message. The intervention arm was subsequently modified to include radio advertising so that the message could be delivered more clearly and directly. This resulted in the following three distinct intervention groups: WOM advertisement of both pOBU and ANC (Intervention A), WOM advertisement of pOBU and WOM + radio advertisement of ANC (Intervention B), and WOM + radio advertisement of both pOBU and ANC (Intervention C). The radio message in Intervention C included the words "You will be able to see a picture of your baby".

All women attending clinic were offered pOBU delivered by a certified Ugandan ultrasound technician using single Nanomaxx unit with a C60n/8-5 MHz (11-mm broadband curved array) probe. Patients rotated through an ANC clinic that was based on the WHO guidelines for high quality ANC5 as well as the WHO four-pronged approach of elimination of mother to child transmission of HIV (EMTCT).

Women received pre- and post-test counseling and rapid testing for HIV. Those who were positive were enrolled into the National HIV program and started on antiretroviral therapy as per national guidelines. Women were also offered intermittent presumptive therapy for malaria, rapid treponemal testing and treatment for syphilis, hepatitis B screening and syndromic management of sexually transmitted infections. Iron and folate supplementation was provided to all women. Any woman in active labour or with a critically low hemoglobin was transported to hospital by ambulance. Any woman with abnormal findings on ultrasound was referred for obstetric specialty follow up. All women were encouraged to deliver at a local HCF.

Survey Women were questioned regarding their experiences and attitudes towards ANC and intentions to utilize a HFC both on entrance (before being debriefed regarding the availability of ultrasound) and after receiving the pOBU results. This was performed with the assistance of a bilingual Ugandan midwife. Data was collected using standardized electronic patient entrance surveys. The forms captured patient demographic and socioeconomic data. Patients were also asked if they were aware of the availability of ultrasound prior to arrival.

Outcomes The primary study outcome was the rate ratio (RR) of total ANC clinic attendance between the intervention groups and control group. Secondary outcomes included A) the RR of attendance by women who had previously used a TBA, B) the RR of attendance by women who had not yet attended ANC, and C) the RR of total attendance between the three interventions.

Statistical Analysis Sub-counties were chosen as the unit of allocation and number of women accessing ANC in each sub-county as the unit of analysis.

The sample size calculation performed a priori was not utilized for this study as the design changed during implementation for reasons specified previously. We performed a post-hoc power calculation. We assumed that the distribution of pregnant women attending ANC was Poisson distributed. We assumed that the number of pregnant women in each community was equal (i.e. we assumed equal offsets for control and intervention arms). We assumed that over-dispersion is not present when conducting the power calculation (i.e. we assumed the Poisson mean is equal to the Poisson variance). Our goal was to test whether the ratio of the Poisson rates was equal to 1 (i.e. the rate of women attending ANC was equal in the control and intervention arms). Assuming a rate ratio of 2, we required 25 women attending ANC in the control arm and 50 women attending ANC in the intervention arm to achieve 80% power to reject the null hypothesis of equal rates of attendance. Assuming a rate ratio of 3, we required 10 women attending ANC in the control arm and 30 women attending ANC in the intervention arm to achieve 80% power to reject the null hypothesis of equal rates of attendance.

Demographic data was summarized using simple descriptive statistics. We computed rates of ANC uptake, first ANC use and ANC uptake due to pOBU, respectively, and all at the cluster level. The count of the number of women attending ANC, for each specific outcome, formed the numerator of the rate. The ideal denominator for the rate calculation would be the number of women who were aware that they were pregnant during the study period. This denominator was unavailable so we used the number of women attending first ANC in 2013-2014 through government run clinics as a proxy. We expressed all rates per 1,000 women. Using Poisson regression, and Pearson's correction factor for over-dispersion, we tested whether the ratio of rates in the control and intervention arms were equal.

We compared the estimated rates in each intervention group with the control group and also in each intervention group with other intervention groups (we computed all possible pair-wise rate ratios between trial arms). We chose to reject the null hypothesis of equal rates of ANC uptake at a 5% alpha level. All statistical analyses were conducted using SAS version 9.4 (Cary, North Carolina). Since the outcomes reported were at the health facility (cluster) level, no further special analyses to account for clustering were conducted.

Role of the Funding Source The funding source of this study was the Canadian not for profit corporation Bridge to Health Medical and Dental (BTH). BTH is primarily funded through unrestricted donations from Canadian corporations (such as Cole Engineering, Lebovic Enterprises and other smaller donors), Canadian Rotary Clubs, and small private donors. None of the donors had any conflicts of interest. None of the Canadian investigators received any personal compensation for their work on this project. The organization has no proprietary holdings on the technology used in this study nor does it, or its investigators, receive any financial compensation for sales of portable ultrasound technology. Some compensation for time spent was provided by BTH to the Ugandan research team.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be residents of the Kabale Region
* All pregnant women aged 18 and above who present to one of the antenatal care clinics

Exclusion Criteria:

* Pregnant women under the age of consent (under 18 years); and any males or non-pregnant females who attend the health camps will be excluded from the study.*

  * All participants excluded from the study will still be offered free medical and dental care as part of a mobile free medical/dental clinic that will be offered in the same community at the same time but in a neighbouring location. For pregnant women under the age of 18, free obstetric ultrasound will also be offered.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Total attendance to antenatal care clinic | 9 days
  The primary outcome in this study was attendance to antenatal care clinic in each sub-county

SECONDARY OUTCOMES:
Attendance to antenatal care clinic by women who had previously seen a traditional healer/birth attendant | 9 days
Attendance to antenatal care clinic by women who had not previously received antenatal care services in their current pregnancy | 9 days
Attendance to antenatal care clinic specifically because of portable obstetric ultrasound | 9 days